CLINICAL TRIAL: NCT05997212
Title: Effect of Repetitive Transcranial Magnetic Stimulation on the Executive Function in Alcohol Use Disorder
Brief Title: Effect of Repetitive TMS on Executive Function in Alcohol Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Eduardo Adrian Garza Villarreal, Assistant Professor, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101.H
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder
Keywords: mri; rtms; tms; repetitive transcranial magnetic stimulation; mexico; magnetic resonance imaging; executive function
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Single-blind randomize clincial trial with parallel groups.
Who Masked: Participant
Masking Description: Single blind. The participants will be the only ones blinded. For placebo or sham we are using vertex as the non-clinical target.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS frequency at 10 Hz (Experimental): The intervention will be Repetitive Transcranial Magnetic Stimulation. Each patient will receive treatment stimulation in the left dorsolateral prefrontal cortex (lDLPFC) with a frequency of 10 Hz, that includes 2 sessions per day for 20 consecutive business days for 4 weeks. Each session will consist of the application of rTMS at a frequency of 10 Hz, to 100% of the motor threshold. The lDLPFC target will be determined using their resting state functional connectivity between anterior cingulate cortex and lDLPFC. Our algorithm performs a calculation of the individual localization of the participant's lDLPFC, which will be used for the whole study in that particular participant.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS frequency at 10 Hz (Sham Comparator): The intervention will be Repetitive Transcranial Magnetic Stimulation (Sham). For this patients the coil will be located on the vertex. Each patient will receive sham stimulation with a frequency of 10 Hz, that includes 2 sessions per day for 20 consecutive business days for 4 weeks. Each session will consist of the application of rTMS at a frequency of 10 Hz, to 100% of the motor threshold. The lDLPFC target will be determined using their resting state functional connectivity between anterior cingulate cortex and lDLPFC. Our algorithm performs a calculation of the individual localization of the participant's lDLPFC, which will be used for the whole study in that particular participant.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (Sham)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — The investigators will use a Magstim Rapid 2 stimulator, Airfilled coil (AFC), 8 shape (magnetic field of 0.8 Teslas, 3Kg, pulse 0.5 ms)
  Each patient will receive high frequency 10 Hz stimulation at 100% of motor threshold over the dorsolateral prefrontal cortex (DLPFC) at 1500 pulses per session with 30 trains of 5 seconds and 0.5 ms stimuli and an inter-train distance of 15 seconds. In 2 daily sessions 4 days a week for 4 weeks.
  Arms: Active rTMS frequency at 10 Hz
Device: Repetitive Transcranial Magnetic Stimulation (Sham) — The investigators will use a Magstim Rapid 2 stimulator, Airfilled coil (AFC), 8 shape (magnetic field of 0.8 Teslas, 3Kg, pulse 0.5 ms)
  Each patient will receive consistent treatment in 2 sessions a day for 20 consecutive business days for 4 weeks. The coil will be placed on the vertex target location.
  Arms: Sham rTMS frequency at 10 Hz

SUMMARY:
Alcohol Use Disorder (AUD) is a major public health problem that affects the physical, social, family, and mental integrity of the sufferer. Behavioral self-regulation is compromised in AUD, and a benefit has been reported with the application of repetitive transcranial magnetic stimulation and emotional self-regulation. The aim of this study is to investigate the efficacy of high-frequency rTMS to improve executive functions in patients in abstinence from AUD.

DETAILED DESCRIPTION:
It is proposed that individuals predisposed to developing alcohol use disorder (AUD) exhibit alterations in executive functions, resulting from maladaptive cellular homeostatic processes and neuronal circuits activated by substance use. These alterations persist even after substance withdrawal (Nestler & Aghajanian, 1997). As a multifactorial disorder, AUD has been linked to family history of alcohol use (Khemiri et al., 2020; Peterson et al., 1990; Tarter et al., 1989) and individual traits such as poor cognitive test performance relative to controls (Shnitko et al., 2018; Goudriaan et al., 2011), which may predict heavy alcohol consumption or AUD development.

These executive dysfunctions manifest as persistent negative behaviors that impede adaptive learning and reduced activation of the executive control network, both of which correlate with AUD severity (Mayhugh et al., 2014). Cognitive flexibility, a key executive function, enables adaptive adjustment of thoughts and behaviors in response to environmental demands (Uddin, 2021). Impaired cognitive flexibility is associated with AUD persistence and severity (Stalnaker et al., 2008), though recovery is observed after prolonged abstinence (Rourke & Grant, 1999). Thus, cognitive flexibility may serve as a promising treatment biomarker.

McLellan et al. (2000) report that 40-60% of AUD patients relapse within the first year post-treatment, while at least 60% relapse within six months (Durazzo & Meyerhoff, 2017; Kirshenbaum et al., 2009; Maisto et al., 2006a; Meyerhoff & Durazzo, 2010). Given these challenges, non-invasive neuromodulation techniques like repetitive transcranial magnetic stimulation (rTMS) have emerged as adjunct therapies to standard treatments (Diana et al., 2017). For example, Addolorato et al. (2017) applied high-frequency (10 Hz) rTMS to the dorsolateral prefrontal cortex (DLPFC) in AUD patients and observed reduced alcohol consumption and increased abstinent days. Similarly, Del Felice et al. (2016) found that left DLPFC stimulation enhanced inhibitory control, selective attention, and mood in active alcohol users.

Stimulating the DLPFC, a hub of the executive control network, may enhance its functional connectivity and improve cognitive flexibility in AUD patients. These effects align with findings that rTMS bolsters inhibitory control and attention (Del Felice et al., 2016; Diana et al., 2017). To explore this further, we propose a longitudinal study assessing cognitive/behavioral traits in AUD patients that may contribute to disorder development. We will also evaluate rTMS effects using neuropsychological tools and MRI to measure structural/functional brain changes.

This study aims to investigate the short- and long-term clinical and cognitive effects of 10 Hz rTMS applied to the left DLPFC in abstinent AUD patients, alongside associated neurostructural and functional connectivity changes. Abstinent AUD patients will receive daily rTMS for four weeks. Clinical outcomes will be tracked for six months, with cognitive, structural, and functional connectivity measurements taken at baseline, post-intervention (4 weeks), and follow-up (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Men and women of 25 to 59 years old
* The reading level of at least 6th grade of primary (equivalent to fifth grade of elementary school).
* Alcohol users with and AUDIT ≥ 20 puntos
* Abstinence from alcohol consumption from 8 weeks to 5 years, with CIWA-Ar scale scores ≤ 9 points.
* No disabling neuropsychiatric conditions (i.e. Schizophrenia)
* No substance use disorders except alcohol and nicotine.
* BrAC (Breath Alcohol) = 0.00 mg/dl in each of the assessments.
* No traces of alcohol consumption using urine test strips.
* No contraindications for TMS therapy.

Exclusion Criteria:

* Individuals with symptoms of severe agitation or who are unable to cooperate in the study
* History of epilepsy
* Sudden onset of stroke, focal neurological findings such as hemiparesis, sensory loss, visual field deficits and lack of coordination.
* Seizures or gait disturbances
* History of severe psychiatric disorders.
* Alterations in a conventional electroencephalogram.
* Pacemakers or intracranial metallic objects.

Elimination criteria

* At the subject's request
* The presence of adverse incidents that deteriorate the subject's health and would limit continuation of rTMS treatment.
* Exacerbation of cognitive or behavioral symptoms during treatment.

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Wisconsin Card Sorting Task | Baseline, 4 weeks
  Measured by Wisconsin Card Sorting Task (WCST) to evaluate cognitive flexibility
Change STROOP effect | Baseline, 4 weeks
  Measured by STROOP test to evaluate control inhibition
Change Visoespatial Memory | Baseline, 4 weeks
  Measured by Visoespatial Memory test to evaluate visoespatial memory

SECONDARY OUTCOMES:
Change in Taskswitching Task Switch cost | Baseline, 4 weeks
  Measured by Taskswitching task to evaluate cognitive flexibility
Change in Flanker Task Flanker Efect | Baseline, 4 weeks
  Measured by Flanker task to evaluate control inhibition
Change in Nback Task accuracy | Baseline, 4 weeks
  Measured by Nback task to evaluate working memory
Change in Alcohol Craving (VAS) | Baseline, 4 weeks, 6 months
  The craving will be measured using a 100 mm visual analogue scales
Changes in psychopathological symptoms | Baseline, 4 weeks, 6 months
  Measured by the Symptoms Questionnaire 90 (SCL-90)
Changes in WHODAS score | Baseline, 4 weeks, 6 months
  Measured by Disability Assessment Schedule (WHODAS)
Changes in Anxiety | Baseline, 4 weeks, 6 months
  Measured by Hamilton Anxiety Rating Scale (HARS)
Changes in Depression | Baseline, 4 weeks, 6 months
  Measured by Hamilton Depression Rating Scale (HDRS)
Changes in functional connectivity | Baseline, 4 weeks
  Functional connectivity of the dorsolateral prefrontal with the anterior cingulate cortex, measured with fMRI defined by the temporal correlation in the blood-oxygen-level-dependent signals of the regions. Higher correlations indicate stronger functional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo A Garza-Villarreal, MD, PhD, Principal Investigator — Universidad Nacional Autonoma de Mexico
Locations (1):
- Unidad de Resonancia Magnética, Querétaro City, Querétaro, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All clinical and MRI data will be shared with each patient's written consent. Identification information will not be shared, only the RID, and all MRI structural data will be defaced prior to sharing. MRI data will be uploaded to Open Neuro while the clinical data will be uploaded to Zenodo.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be shared once the study is finished and published, aproximately in 2027
Access Criteria: open access